CLINICAL TRIAL: NCT04804332
Title: Removal of Intrauterine Retained Products of Conception (RPOC) After Miscarriage Guided by Hysteroscopy Trial. A Randomized Controlled Trial.
Acronym: RIGHT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-08856
Record Dates: First submitted 2021-03-08; First posted 2021-03-18 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Retained Products of Conception
Keywords: Retained Products of Conception; placental remnants; hysteroscopy; expectant management; fertility
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Intervention Model Description: Design : RCT
  * Multicenter
  * Randomized controlled
  * Parallel group design
  * Superiority trial
  * Non-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPECTANT MANAGEMENT (Experimental): No treatment will be offered.
  Interventions: Other: Expectant management
- OPERATIVE HYSTEROSCOPY (Experimental): Operative hysteroscopy using hysteroscopic morcellation (TruClearTM Hysteroscopic Tissue Removal System (Medtronic, Minneapolis, MN, USA)) is performed.
  Interventions: Procedure: Operative hysteroscopy

INTERVENTIONS:
Procedure: Operative hysteroscopy — Operative hysteroscopy is performed without or under local, regional or general anesthesia according to the local protocol preferably within 2 to 3 weeks after randomization. In case of highly vascularized RPOC, a repeat sonogram is performed 2 to 4 weeks after randomization to check for persistence of vascularity and to optimize operative timing. Operative hysteroscopy is then performed within 2 to 3 weeks after the repeat sonogram. Removal of the RPOC is performed by an experienced gynecologist using hysteroscopic morcellation (TruClearTM Hysteroscopic Tissue Removal System (Medtronic, Minneapolis, MN, USA)) and according to the local protocol.
  Arms: OPERATIVE HYSTEROSCOPY
Other: Expectant management — No treatment will be offered. Patients will be given telephone numbers to contact a doctor. In case of severe complaints, defined as heavy uterine bleeding and/or severe abdominal pain, not responding to conservative treatment, an emergency curettage or operative hysteroscopy may be performed.
  Arms: EXPECTANT MANAGEMENT

SUMMARY:
Rationale: Elective immediate dilation and curettage (D&C) for miscarriage is associated with the occurrence of intrauterine adhesions (IUA). IUAs may be associated with subsequent subfertility and premature birth. Recent studies have shown that in women with miscarriage, medical treatment (misoprostol/mifepristone) is an effective alternative for curettage. A problem with medication and expectant management is that after initial treatment, sonographic findings during follow-up frequently show incomplete evacuation of uterine retained products of conception (RPOC), which often lead to additional interventions or expectant time-consuming management limiting the benefits of medical treatment.

Objective: To assess, in women with a wish for immediate future pregnancy and RPOC after non-surgical management of a miscarriage, as diagnosed with sonography, the effects of operative hysteroscopy versus expectant management.

Study design: Multicenter randomized clinical trial. Study population: Patients after non-surgical management of a miscarriage with sonographic evidence of RPOC at the follow-up visit 6 weeks after initial treatment and wish for immediate (within 6 months) future pregnancy.

Intervention: operative hysteroscopy versus expectant management. Main study parameters/endpoints: The primary outcome is time to next pregnancy, as substantiated by a positive urinary or serum hCG test. Secondary outcomes are Quality of Life (QOL) scores assessed with the SF-36, HADS and EQ-5D-5L, the need for additional and/or unscheduled treatments and/or visits and complications. Furthermore, data on the course of pregnancy - including miscarriage, ectopic pregnancy and live birth - are documented in those women who have an ongoing pregnancy after randomization during the study follow up period. In addition, iMTA PCQ questionnaires and health-costs are measured in all patients to perform a cost-effectiveness analysis.

A total of 244 (122 per arm) women will be sufficient to answer the questions on the primary endpoint.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Women participating in the study will be asked to fill out questionnaires at baseline, 8 weeks and 6 months after randomization. We don not expect specific risks as a result of either the intervention or expectant management.

DETAILED DESCRIPTION:
Design : RCT

* Multicenter
* Randomized controlled
* Parallel group design
* Superiority trial
* Non-blinded

Primary Objective

To compare the effectiveness in terms of time to next pregnancy between operative hysteroscopy and expectant management in patients with sonographic evidence of RPOC after primary non-surgical management of miscarriage.

Secondary Objectives

1. Effectiveness objectives

   To compare the effectiveness between operative hysteroscopy and expectant management with respect to:
   * Generic quality of life (QOL) (as measured by SF-36, HADS (Hospital Anxiety and Depression Scale)) and EQ-5D-5L 6 months after randomization
   * Course of pregnancy in those women who have an ongoing pregnancy after randomization during the study follow-up period (including miscarriage, ectopic pregnancy and live birth)
2. Safety objectives

   To compare the safety between operative hysteroscopy and expectant management with respect to:
   * Necessity for additional treatment
   * Out-of-protocol/unscheduled visits to the outpatient clinic or general practitioner
   * Complications
3. Cost-effectiveness objectives To compare the health related costs between operative hysteroscopy and expectant management.

ELIGIBILITY:
Inclusion Criteria:

* Patients after first trimester miscarriage treated non-surgically with sonographic evidence for the presence of RPOC at follow-up visit after 6 weeks (± 1 week) who have an immediate future pregnancy wish and are willing to give informed consent.

Exclusion Criteria:

* Women aged below 18 years
* Women aged over 39 years
* Women not wanting to achieve pregnancy within the first 6 months after non-surgical treatment for miscarriage
* Women with a history of repeated miscarriage defined as 3 or more consecutive pregnancy losses before 20 weeks of pregnancy duration
* Women with untreated and/or untreatable subfertility
* Women presenting with severe uterine bleeding, defined as uterine bleeding that needs acute intervention on medical grounds
* Women presenting with severe abdominal pain, defined as abdominal pain that needs acute intervention on medical grounds
* Women with fever (> 38.5° Celsius) or sepsis requiring antibiotic treatment. For the definition of 'sepsis' we refer to the Third International Consensus definitions for Sepsis and Septic Shock (Singer 2016)
* Women with a contraindication for (office) operative hysteroscopy
* Women with a failed non-surgical management for miscarriage, as substantiated by the sonographic finding of an intact gestational sac still in situ
* Women with a congenital uterine anomaly
* Known cervical stenosis making safe uterine access impossible
* Visual or pathological (e.g. on biopsy) evidence of malignancy

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 244 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to next pregnancy | up to 3 years after the start of the trial
  The primary endpoint is the time until next pregnancy since randomization, with pregnancy defined as a positive urinary or serum hCG test. Patients are asked to contact the study team in case of pregnancy. If a participant has failed to contact the center, pregnancy will be asked at same time as the questionnaires and then once every 6 months as well as at the end of the study by telephone contact or e-mail.

SECONDARY OUTCOMES:
Quality Of Life (QOL) | at baseline, 8 weeks after randomization and 6 months after randomization
  measured by SF-36
Quality Of Life (QOL) | at baseline, 8 weeks after randomization and 6 months after randomization
  measured by HADS (Hospital Anxiety and Depression Scale)
Quality Of Life (QOL) | at baseline, 8 weeks after randomization and 6 months after randomization
  measured by EQ-5D-5L
Course of pregnancy | up to 3 years after the start of the trial
  Course of pregnancy in those women who have an ongoing pregnancy after randomization during the study follow-up period (including miscarriage, ectopic pregnancy and live birth):
  * Time to conception, defined as the time from randomization to the date of conception retrospectively determined based on the crown-rump length measurement (CRL) by a first-trimester ultrasound.
  * Clinical pregnancy defined as a pregnancy diagnosed by ultrasonographic visualization of 1 or more gestational sacs or definitive clinical signs of pregnancy, including ectopic pregnancy. Multiple gestational sacs are counted as 1 clinical pregnancy.
  * Live birth, defined as the complete expulsion or extraction from the mother of a product of fertilization, irrespective of the duration of pregnancy, which after such separation breathes or shows any other evidence of life, such as heartbeat, umbilical cord pulsation, or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been
Necessity for additional treatment | until 6 months after randomisation
  Necessity for additional treatment
Out-of-protocol/unscheduled visits | until 6 months after randomisation
  Re-interventions or additional treatment during the first 6 months including type, number and reasons.
  Out-of-protocol visits to the outpatient clinic or general practitioner or hospitalizations including type, number, reasons and duration of hospitalization.
Complications | until 6 months after randomisation
  Heavy uterine bleeding defined as uterine bleeding that needs acute intervention (IV iron administration, tranexamic acid or blood transfusion) on medical grounds
Complications | until 6 months after randomisation
  Severe abdominal pain requiring analgesics or medical intervention, excluding postoperative pain in the first 48 hours after uterine surgery
Complications | until 6 months after randomisation
  Fever (>38.5° Celsius) or sepsis
Complications | until 6 months after randomisation
  - Related to operative hysteroscopy or other surgical treatment
  * uterine perforation
  * postoperative hemorrhage, defined as excessive blood loss estimated or measured as ≥ 500 mL and/or need for blood transfusion
  * severe abdominal pain requiring analgesics excluding postoperative pain in the first 48 hours after hysteroscopic surgery
  * fluid overload (defined as absorption of more than 2500 mL of distention medium with clinical consequences for the patient)
  * electrolyte disturbances requiring treatment
  * gas embolism
Health related costs | until 6 months after randomisation
  the EQ-5D-5L and health-related costs based on physician visits, hospitalizations and emergency room visits are measured

CONTACTS AND LOCATIONS:
Overall Officials: Tjalina Hamerlynck, MD PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No